CLINICAL TRIAL: NCT00348907
Title: Evaluation of the Efficacy of the Thermal Cure in the Prevention of the Post-Thrombotic Syndrome After a Deep Venous Thrombosis of Lower Limbs.
Brief Title: EVENT: Hydrotherapy and Deep Venous Thrombosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: decision to stop the study because of enrollment difficulties.
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCIC 05 45
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Pain; Deep Venous Thrombosis
Keywords: doppler; CIVIQ quality of life; Hydrotherapy; anticoagulants
MeSH Terms: conditions — Pain; Venous Thrombosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): immediate thermal cure (1st year)
  Interventions: Drug: thermal cure
- 2 (Sham Comparator): late thermal cure (2 years)
  Interventions: Drug: late thermal cure

INTERVENTIONS:
Drug: thermal cure — thermal cure of 18 days including movement in swimming pool, mud-bath, shower, massage and thermal steam
  Arms: 1
Drug: late thermal cure — thermal cure of 18 days including movement in swimming pool, mud-bath, shower, massage and thermal steam at 2 years
  Arms: 2

SUMMARY:
The main objective of this study is to demonstrate that hydrotherapy in a specific place can reduce the risk of post-thrombotic syndrome.

DETAILED DESCRIPTION:
Venous thrombo-embolic disease (VTED) is a frequent pathology. The incidence is about 5 to 20 cases for 10000 persons each year, in a general population. The immediate risk is the pulmonary embolism potentially fatal. So, it justifies all the works in clinical research during the last years. Those studies allow many progresses, diagnostic and therapeutic, for the immediate undertaking of the patients. Despite that, VTED is a major problem of public health and the diminution of the mortality lied to VTED is one of the objectives of the French law relative to the politics of Public Health (August 2004). At more long-term, the post-thrombotic syndrome lead to an incapacitating pathology, which requires many cares. The frequency of the post-thrombotic syndrome is evaluated between 25 and 60% at middle-term (1 or 2 years). It depends of the studies and of the clinical primary end-points or vascular explorations. Rehabilitation has never been validated in this indication by studies with a correct methodology.

Deep venous thrombosis (not in acute phase) is recognized as an indication for about 10 spa in France. But the specific or global benefit of this water cure is not clearly and scientifically proved. The importance of the venous pump of the calf and of the hydrostatic pressure in the physiopathology of the post-thrombotic syndrome make natural the use of balneotherapy for the prevention of this pathology for patients with severe deep venous thrombosis of lower limbs (proximal and obstruent). The venous thermal techniques have well-defined physiopathological targets. The haemodynamic and microcirculatory effects of some of them have been proved. The high degree of satisfaction of the patients that benefit from phlebological water cure every year in France indirectly shows the benefits that they feel. In those indications, prevention of the post-thrombotic syndrome is one of the well-recognize by the medical profession. For all that, there was not really validation of this indication with an acceptable methodology for the canons of the modern medicine. That is the reason why we undertake this randomized, single-blind controlled study with for main objective to demonstrate that hydrotherapy in a specific place can reduce the risk of post-thrombotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* both sexes;
* 18 years old and more;
* clinical indication of thermal cure (first phase of deep venous thrombosis authenticated by unilateral venous echo-doppler
* curative anticoagulant treatment more than 3 month;
* oedema and/or spontaneous pain with functional discomfort;
* available for a thermal cure during 18 days and a follow-up period of 36 month;
* voluntary to participate to the study, informed consent form signed after appropriate information;
* affiliation to the social security system or equivalent;
* no previous participation to a thermal cure (in the indication of phlebology)

Exclusion Criteria:

* isolate distal thrombosis;
* asymptomatic thrombosis;
* cutaneous ulcer of lower limb;
* refusal to consent;
* refusal to benefit of thermal cure;
* contra-indication to hydrotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Presence at 1 year of a severe post-thrombotic syndrome clinically defined. | 1 year

SECONDARY OUTCOMES:
Post-thrombotic syndrome at 2 years; | 2 years
Quality of life: CIVIQ Scale; | inclusion, 1, 2 years before and after thermal cure
Intensity of the symptoms of venous insufficiency auto evaluation by patient | monthly
Deep venous reflux (evaluated by echo-doppler); | inclusion, 1 and 2 years
Persistence of a residual thrombus (echo-doppler); | inclusion, 1 and 2 years
Correlation between clinical evolution and echo-doppler evolution of the venous after-effects; | 1 year
Benefit of a late cure at 2 years. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François POIRAULT, Dr, Principal Investigator
Locations (27):
- France (27):
  - Etablissement thermal, Argelès-Gazost
  - Etablissement thermal, Bagnoles-de-l'Orne
  - Etablissement thermal, Barbotan-les-Thermes
  - L'avenue, Dax
  - Sarrailh, Dax
  - Le Splendid, Dax
  - Les thermes, Dax
  - Le miradour, Dax
  - Les arènes, Dax
  - Bérot, Dax
  - Les écureuils, Dax
  - Dax thermal, Dax
  - Foch, Dax
  - Borda, Dax
  - Saint-Pierre, Dax
  - Le Grand Hôtel, Dax
  - Le Regina, Dax
  - Etablissement thermal, Évian-les-Bains
  - Domaine d'heurteboise, Jonzac
  - Etablissement thermal, La Léchère
  - Etablissement thermal, Luxeuil-les-Bains
  - Etablissement thermal, Luz-Saint-Sauveur
  - Etablissement thermal, Rochefort
  - Caliceo, Saint-Paul-lès-Dax
  - Christus, Saint-Paul-lès-Dax
  - Chênes, Saint-Paul-lès-Dax
  - Etablissmeent thermal, Saubusse-les-bains

REFERENCES:
- [Background] Prandoni P, Lensing AW, Cogo A, Cuppini S, Villalta S, Carta M, Cattelan AM, Polistena P, Bernardi E, Prins MH. The long-term clinical course of acute deep venous thrombosis. Ann Intern Med. 1996 Jul 1;125(1):1-7. doi: 10.7326/0003-4819-125-1-199607010-00001. PMID 8644983
- [Background] Kahn SR, Kearon C, Julian JA, Mackinnon B, Kovacs MJ, Wells P, Crowther MA, Anderson DR, Van Nguyen P, Demers C, Solymoss S, Kassis J, Geerts W, Rodger M, Hambleton J, Ginsberg JS; Extended Low-intensity Anticoagulation for Thrombo-embolism (ELATE) Investigators. Predictors of the post-thrombotic syndrome during long-term treatment of proximal deep vein thrombosis. J Thromb Haemost. 2005 Apr;3(4):718-23. doi: 10.1111/j.1538-7836.2005.01216.x. Epub 2005 Feb 23. PMID 15733061
- [Background] Labropoulos N, Leon LR Jr. Duplex evaluation of venous insufficiency. Semin Vasc Surg. 2005 Mar;18(1):5-9. doi: 10.1053/j.semvascsurg.2004.12.002. PMID 15791546
- [Background] Asbeutah AM, Riha AZ, Cameron JD, McGrath BP. Reproducibility of duplex ultrasonography and air plethysmography used for the evaluation of chronic venous insufficiency. J Ultrasound Med. 2005 Apr;24(4):475-82. doi: 10.7863/jum.2005.24.4.475. PMID 15784766
- [Background] Launois R, Reboul-Marty J, Henry B. Construction and validation of a quality of life questionnaire in chronic lower limb venous insufficiency (CIVIQ). Qual Life Res. 1996 Dec;5(6):539-54. doi: 10.1007/BF00439228. PMID 8993100